CLINICAL TRIAL: NCT04517019
Title: Randomisierte Studie Zum Nutzen Eines Fitnesstracker Basierten Aktivitätstrainings während Einer Strahlentherapeutischen Behandlung (OnkoFit II Studie)
Brief Title: Randomised Trial Evaluating the Benefit of a Fitness Tracker Based Workout During Radiotherapy
Acronym: OnkoFit II
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Dr. Cihan Gani, Senior Physician, University Hospital Tuebingen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: OnkoFit II
Record Dates: First submitted 2020-08-13; First posted 2020-08-18 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Bronchial Carcinoma; Esophageal Carcinoma; Tumor of the Brain; Head and Neck Cancer; Pancreas Cancer; Sarcoma; Cervix Uteri Cancer
Keywords: Fatigue; Activity tracker; Radiotherapy; Exercise
MeSH Terms: conditions — Carcinoma, Bronchogenic; Esophageal Neoplasms; Brain Neoplasms; Head and Neck Neoplasms; Pancreatic Neoplasms; Sarcoma; Uterine Cervical Neoplasms; Fatigue; Motor Activity | interventions — Exercise Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm A (Tracker/daily step-count suggestion) (Experimental): Patients receive a fitness tracker, a booklet "Physical training, exercise and cancer" and an in-person briefing on physical activity during cancer therapy. We suggest a daily step-count which should improve the patients phyiscal activity during radiotherapy of breast cancer. Patients receive weekly feedback and a new goal with the aim to reach a total of 6000 daily steps, which should be then maintained during radiotherapy.
  Interventions: Device: Fitness tracker based activity training for Arm A and B. Booklet "physical training, exercise and cancer" and an introduction about physical activity during cancer therapy for Arm A, B, C
- Arm B (Tracker/no daily step-count suggestion) (Experimental): Patients receive a fitness tracker, a booklet "Physical training, exercise and cancer" and an in-person briefing on physical activity during cancer therapy.
  The patients self-document their daily step count during radiotherapy, there will be no recommendation for the daily count of steps.
  Interventions: Device: Fitness tracker based activity training for Arm A and B. Booklet "physical training, exercise and cancer" and an introduction about physical activity during cancer therapy for Arm A, B, C
- Arm C (no activity tracker) (No Intervention): Patients receive a booklet "Physical training, exercise and cancer" and an in-person briefing on physical activity during cancer therapy. A fitness tracker will not be provided.

INTERVENTIONS:
Device: Fitness tracker based activity training for Arm A and B. Booklet "physical training, exercise and cancer" and an introduction about physical activity during cancer therapy for Arm A, B, C — Patients receive a fitness tracker, a booklet "Physical training, exercise and cancer" and an in-person briefing about physical activity during cancer therapy. With offered guidelines for the daily step counts patients should improve their physical activity during radiotherapy of breast cancer. A weekly feedback and a new goal for the next week will be provided until the individual patient reaches a daily activity of 6000 steps. The setting will be to maintain to this daily activity of 6000 steps during radiotherapy.
  Arms: Arm A (Tracker/daily step-count suggestion); Arm B (Tracker/no daily step-count suggestion)

SUMMARY:
Evaluation of the impact of an activity tracker based fitness programme on the Qualitiy of Life after oncological therapy.

DETAILED DESCRIPTION:
This monocentric, three-arm, randomized, controlled clinical trial evaluates the effect of an activity tracker based exercise program in cancer patients on the Quality of life after oncological therapy. Quality of Life and the intensity of fatigue will be documented with the FACT-G total score of the FACIT Questionnaire six months after completion of radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Capacity for consent
* Minimum age 18
* Presence of one of the following tumor diseases: Bronchial Carcinoma, Esophageal Carcinoma, Tumor of the Brain, Head and Neck Cancer, Pancreas Cancer, Sarcoma Cervix Uteri Cancer
* ECOG 0-2
* Indication for a radiotherapy or a radiochemotherapy with an intended treatment time of minimum 4 weeks (definitive/adjuvant/neoadjuvant)

Exclusion Criteria:

* Participation in any other interventional study
* Radiotherapy of Breast cancer
* Pregnancy
* Contraindication against physical activity/sport and others
* Severe cardiovascular pre-existing conditions (after myocardial infarction, apoplexy in the last 6 months, congestive heart failure NYHA > I°)
* preexisting diseases with are relevantly accompanied by a limited mobility in patients (e.g. paraparesis of the lower limbs)
* ECOG Status 3-4
* prior use of activity trackers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the impact of an Activity tracker based Fitness programme on the Qualitiy of Life after oncological Therapy | 6 Months after completion of adjuvant radiotherapy
  This endpoint will be evaluated by the FACT-G (Functional Assessment of Cancer Therapy - General) total scores of the FACIT (Functional Assessment of Chronic Illness Therapy) questionnaire (physical well-being values 0-28, 28 worse outcome; social/family well-being values 0-28, 28 better outcome; emotional well-being values 0-24, 24 worse outcome; functional well-being values 0-28, 28 better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Cihan Gani, MD, PD, Principal Investigator — University Hospital Tübingen
Locations (1):
- University Hospital Tübingen, Tübingen, Baden-Wurttemberg, Germany

REFERENCES:
- [Derived] Hauth F, Gehler B, Niess AM, Fischer K, Toepell A, Heinrich V, Roesel I, Peter A, Renovanz M, Hartkopf A, Stengel A, Zips D, Gani C. An Activity Tracker-Guided Physical Activity Program for Patients Undergoing Radiotherapy: Protocol for a Prospective Phase III Trial (OnkoFit I and II Trials). JMIR Res Protoc. 2021 Sep 22;10(9):e28524. doi: 10.2196/28524. PMID 34550079